CLINICAL TRIAL: NCT05550623
Title: Pneumatic Tourniquet Versus no Tourniquet in Transfemoral Amputation - A Randomized Controlled Trial
Brief Title: Pneumatic Tourniquet Versus no Tourniquet in Transfemoral Amputation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anna Trier Heiberg Brix, Medical Doctor, PhD Student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2202766
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Amputation; Blood Loss
Keywords: Tourniquet; Major Lower Extremity Amputation; Transfemoral Amputation; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Tourniquets

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, two-arm, blinded trial. Superiority-design Allocation 1:1 Eligible patients will be randomized to transfemoral surgery with or without the application of a sterile pneumatic tourniquet.
Who Masked: Participant
Masking Description: Blinding Participants and staff not attendant in the room will be blinded. The use of tourniquet will not be visible in the patient records but recorded directly in the REDCap Database. A standard phrase to describe the surgical procedure will be used in the patient record. Deviations and adverse events will be described. Participants will be able to be informed by the procedure after 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transfemoral amputation performed with tourniquet application (Experimental): Group 1:Randomized to procedure with Tourniquet application Sterile wash to groin and placement of sterile tourniquet. The amputation level approximately 10-15 cm above the upper edge of patella is marked and the anterior and posterior flaps are measured and drawn out.
  The leg is lifted, and the tourniquet is inflated. The pressure is set to 250 mmHg. Starting time is noted. Incision through skin, fascia and musculature. The femoral vessels are clamped, cut and ligated. With an oscillating saw the femoral bone is cut, and the leg can be removed The tourniquet is deflated. Tourniquet time is noted. Rest of procedure as listed in arm2
  Weight of the leg is noted. Weight of surgical swabs is noted, to estimate intraoperative blood loss.
  Interventions: Device: Tourniquet
- Transfemoral amputation performed without tourniquet application (No Intervention): Group 2: Randomized to procedure without Tourniquet The amputation level approximately 10-15 cm above the upper edge of patella is marked and the anterior and posterior flaps are measured and drawn out. Incision through skin, fascia and musculature. The femoral vessels are clamped, cut and ligated. With an oscillating saw the femoral bone is cut, and the leg can be removed.
  The edge of the femoral bone is rasped smooth. A myodesis is performed, attaching the adductor muscle to the end of the femoral bone. Nervus Ischiadicus is dissected as proximal as possible and protected within a purse string suture to avoid development of neuroma.
  Ligation of bleeding vessels. Fascia and skin is closed with sutures. A soft compression bandage is applied to the stump.
  * Weight of the leg is noted.
  * Weight of surgical swabs is noted, to estimate intraoperative blood loss.

INTERVENTIONS:
Device: Tourniquet — Tourniquet use in transfemoral amputation.
  Arms: Transfemoral amputation performed with tourniquet application

SUMMARY:
Lower extremity amputation patients represent a frail group of patients with extensive comorbidity. The most common indication of amputation is ischemia, infection and concomitant ischemic pain due to underlying chronic disease, especially arteriosclerosis and diabetes.

Prolonged general anesthesia and surgery as well as increased blood loss may result in impaired patient safety. Previous studies have shown total blood loss approx. 1000 mL in transfemoral amputations (TFA). Substantial blood loss during surgery increases the risk of anemic complications and death for this already weakened patient group.

The aim of this randomized controlled trial is to improve patient safety by exploring the possibility of a more precautious surgical procedure for TFA. Hence, investigating the total blood loss and secondary differences in complications after TFA between patients operated with use of pneumatic tourniquet versus no tourniquet. Total blood loss is calculated via Nadlers approach. From a pilot series, sample size was calculated to 124, allocated 1:1 in two groups of 62 participants, to ensure detection of at least 200 mL difference in total blood loss.

The hypothesis is that use of tourniquet will decrease the total blood loss, the amount of blood transfusions, time of surgery and complications related to postoperative anemia without a higher rate of adverse events. The secondary and explorative outcomes are blood transfusions, intraoperative blood loss, length of stay, time of surgery, risk of readmission, risk of re-operation, risk of mortality, complications during admission, quality of life (QoL), prosthesis use and the prosthesis-specific survey Prothesis Evaluation Questionnaire (PEQ). QoL is measured with the validated questionnaire EQ-5D-5L preoperatively, and at 3, 6, and 12 months postoperatively.

The possibility to enhance patient safety is highly relevant, and this trial will aid in establishing evidence-based guidelines for TFA surgery.

DETAILED DESCRIPTION:
Hypothesis The hypothesis is that the use of tourniquet in Transfemoral amputation (TFA) surgery will reduce the total blood loss, the intraoperative blood loss and the need for blood transfusion post-operatively and thereby improve patient safety.

Aim Primary to investigate total blood loss and secondary to investigate differences in complications after TFA surgery between patients operated with use of pneumatic tourniquet versus no tourniquet.

Trial design overview Design: Randomized, prospective, blinded, two-arm, single center trial. Superiority-design. Group 1: Transfemoral amputation performed with tourniquet application Group 2: Transfemoral amputation performed without tourniquet application Population: Patients with indication for primary transfemoral amputation (intact femoral bone). Period: Expected trial inclusion period is October 2022- September 2024. Place: Odense University Hospital (OUH), Odense, Denmark Sample size: 62 in each group, a total of 124 participants inclusive a 20 % buffer.

The flow of TFA patients in the department is approximately 100 patients annually and it will therefore be possible to include the calculated sample size in the time frame available for this trial.

Tourniquet: The tourniquet that is used at OUH is FastAir® distributed and imported by Universal Medical Supplies Aps. Universal Medical Supplies Aps is not a part of this protocol.

This trial is not conducted in collaboration with Universal Medical Supplies Aps. Universal Medical supplies Aps has no right to unpublished study data and is neither financially nor personally involved in this trial. None in the study group is related to Universal Medical Supplies ApS. MDR classification for FastAir® tourniquet: class I, non-invasive device for temporary use.

The FastAir® tourniquet has a CE-certificate. The FastAir® tourniquet will be used according to instructions for use. Tourniquet application for transfemoral amputation at OUH is not standard of care.

Randomizing and database Randomization is performed internet-based using REDCap Randomize, allocation 1:1. The randomization itself takes place in the period 4 weeks prior to surgery to immediately before surgery. The randomization is performed as a block randomization and will be stratified for age (>70 years / ≤70 years) and hemoglobin value pre surgery (>6mmol/L / ≤6 mmol/L). Two stratifies is acceptable for the calculated sample size.

Blinding Participants and staff not attendant in the room will be blinded. The use of tourniquet will not be visible in the patient records but recorded directly in the REDCap Database. A standard phrase to describe the surgical procedure will be used in the patient record. Deviations and adverse events will be described. Participants will be able to be informed by the procedure after 6 months.

Feasibility In a pilot study, feasibility of tourniquet application was assessed. The pilot-study was carried out in the department in May-July 2021. Placement of tourniquet for TFA surgery is generally possible in >90%. The blood tests are not always drawn at third day post surgery, but this will be assessed in the new department algorithm for postoperative care for major lower extremity amputation patients, to ensure correct data collection in this study. The mean application time of the tourniquet was 12,15 minutes (5 minutes -21 minutes).

Sample Size From the pilot series there was observed a mean of 429 ml and standard deviation (SD) of 199 ml in 11 intervention procedures (with tourniquet) and a mean of 730 ml and SD of 446 ml in 12 control procedures (without tourniquet). The calculated blood loss in each group was normally distributed according to quantile-quantile plots (Appendix 1). It is assumed that a mean difference of 200 ml would be lower than any reasonable clinically important difference, and hence chose this as the difference for our sample size calculation.

From this,there was calculated the need of 49 participants in each group for a two-sample t-test fora superiority trial. To take into account for up to 20% drop-out (e.g. due to invalid data/protocol violation/intraoperative mortality/participant wish/investigator indication), it was decided to include 62 participants in each group (49/0,8=61,25). The sample size calculation was performed in Stata/IC 16.1with help from OPEN Statistics,OUH.

Screening log is performed on patients not included, to examine the cause of non-inclusion.

Patients that are not included in this study, no matter of cause, will be offered to participate in a concurrently prospective non-interventional cohort study where the main outcome is health related quality of life before and after surgery. These patients will only receive electronic surveys (in E-boks) regarding quality of life (EQ-5D), disease course, pain, mobility and daily life. This will serve as drop-out analysis. The same baseline data will be recorded on these patients. They will receive the department standard treatment.

Statistical analysis plan The investigators will report descriptive statistics of patient characteristic as mean and standard deviation (SD) for normally distributed, median and interquartile range (IQR) for non-normally distributed, and counts and proportions for categorical characteristics. The investigators will compare the primary outcome (calculated blood loss) by two-sample t-test with unequal variance and report mean and SD for each group as well as the mean difference with a 95% normal confidence interval (CI). The investigators will report the dichotomous secondary and exploratory outcomes as counts and proportions, compare these with chi-squared test (or Fisher's exact test, if any counts are below five) and report odds ratios with 95% CI from crude logistic regression. The investigators will report numerical secondary and exploratory outcomes either as means and SD and compare those by two-sample t-test, if deemed normally distributed by quantile-quantile plots, or otherwise, as medians and IQR and compared by Wilcoxon rank-sum test if not deemed normally distributed. All analyses will be carried out as a superiority design and as intention to treat analysis is performed for all included participants, and p-values below 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Speak and understand Danish and able to give informed consent
* ≥18 years of age
* Indication for first transfemoral amputation (intact femur)

Exclusion Criteria:

* Bilateral amputation in same procedure
* Femoral amputation revision (non-intact femur)
* Malignant disease as main cause of amputation
* Not possible to place tourniquet correctly (surgeon assessment)
* Acute trauma
* Planned surgery with surgeon charged less than second year residents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Total blood loss calculated using Nadler's approach | Day 1- Day3
  To calculate this outcome the following information is needed: gender, weight, height, hemoglobin value before surgery (accepted timespan 4 weeks before surgery to day of surgery), hemoglobin value on the third day post surgery, and the number of blood transfusions (from day of surgery to third postoperative day).

SECONDARY OUTCOMES:
Blood transfusion | Day 1- Day 3
  Transfusions received in the period from the measured hemoglobin preoperatively to the third postoperative day.
Intraoperative blood loss | Day 1
  Estimated value. Measured in surgery as weight difference in surgical swabs and measured suction blood
Length of stay | Day 1 - To discharge or date of death, whichever comes first, with a maxium of 52 weeks
  Length of stay is defined as postoperative nights in hospital, including transfers to other departments/hospitals, until discharge to home or rehabilitation unit.
Complications during admission | Day 1 - To Discharge or date of death, whichever comes first, with a maxium of 52 weeks
  Complications will be grouped using the OrthoSAVES guidelines
Risk of mortality ≤30 days | Day 1 - Day 30
  Data from patient records, combined with data from the CPRregistry
Risk of readmission ≤90 days | Day 1 - Day 90
  Readmission is defined in at least one overnight stay. Readmissions due to planned procedures or obviously unrelated to surgery are not included
Risk of re-operation ≤30 days and ≤90 days | Day 1- Day 90
  Defined as same site surgery, whether amputation at a higher level where the femoral bone shortened or revision of soft-tissue

OTHER OUTCOMES:
Risk of re-operation ≤ 1 year | Day 1 - Day 365
  Defined as same site surgery, whether amputation at a higher level where the femoral bone shortened or revision of soft-tissue. All re-operations in the one-year period after index surgery will be included for analysis.
Risk of mortality ≤ 1 year | Day 1 - Day 365
  Data from patient records, combined with data from the CPRregistry
Prosthesis user ≤ 1 year | Day 1 - Day 365
  The amount of participants that will be prosthesis users in the first year after amputation.
Quality of Life (EQ-D5) | Day 1 - Day 365
  The ED-5Q-5L is a validated survey for measuring HRQoL It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analog scale. The participants will answer EQ-5D electronically before surgery (at booking or at admission to department), 3 months after, 6 months after and 12 months after index TFA surgery. The outcome is reported on a scale of 1-5 where 1 is no problems and 5 is extrem problems.
Prosthesis Evaluation Questionnaire (PEQ) | Day 365
  The Prosthesis Evaluation Questionnaire (PEQ) is translated to Danish and assesses prosthesis related quality of life in nine subscales.
  The Danish validation showed reliability for six subscales and mixed results for the last three subscales. To use this survey prosthesis must be used. According to the Swedish amputation registry mean time from amputation to prosthesis fitting is approx. four to five months for TFA and 2-3 months after Transtibial Amputation (TTA) . PEQ will be answered at 12 months post surgery, for those participants that received prosthesis in the study period. The subscales are Ambulation, Appearance, frustation, Percived response, residual limb health, Social burden, sounds, utility and well being. The score is reported on a VAS scale, as an avarage, of those questions in the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lindberg-Larsen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brix ATH, Nymark T, Schmal H, Lindberg-Larsen M. Pneumatic tourniquet versus no tourniquet in transfemoral amputation - a study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2022 Dec 13;23(1):1088. doi: 10.1186/s12891-022-06000-6. PMID 36514077

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT05550623/SAP_000.pdf